CLINICAL TRIAL: NCT02737813
Title: Cardiac Output Changes During Hyperbaric and Isobaric Bupivacaine in Patients Undergoing Cesarean Section: An Randomization Trials
Brief Title: Cardiac Output Changes During Hyperbaric and Isobaric Bupivacaine in Patients Undergoing Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Marcaine
Record Dates: First submitted 2016-03-23; First posted 2016-04-14 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Output; Hypotension; Anesthesia, Spinal
Keywords: isobaric marcaine; hyperbaric marcaine
MeSH Terms: conditions — Hypotension | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isobaric Marcaine (Experimental): Isobaric Marcaine 2.2 mL for spinal block
  Interventions: Drug: Isobaric marcaine
- Hyperbaric Marcaine (Active Comparator): Hyperbaric Marcaine 2.2 mL for spinal block
  Interventions: Drug: Hyperbaric marcaine

INTERVENTIONS:
Drug: Isobaric marcaine — Isobaric marcaine 2.2 mL for spinal block
  Other Names: bupivacaine
  Arms: Isobaric Marcaine
Drug: Hyperbaric marcaine — Hyperbaric marcaine 2.2 mL for spinal block
  Other Names: bupivacaine
  Arms: Hyperbaric Marcaine

SUMMARY:
Spinal block leads to the reduction of systemic vascular resistance (SVR) which may effect the cardiac output. Ngan Kee et al. has showed that spina block with 0.5% hyperbaric bupivacaine for Cesarean section combined with intravenous infusion norepinephrine had higher cardiac output than those who received phenylephrine

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology classification I - II
* Elective or urgency Cesarean section with spinal block e.g. cephalopelvic disproportion, premature rupture of membrane
* Singleton pregnancy
* Body mass index < 40 kg/m2

Exclusion Criteria:

* Pregnancy <35 weeks gestational age
* Hypertensive disease e.g. gestational hypertension, chronic hypertension, preeclampsia
* History of allergy to the study drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Change of cardiac output (L/min) after spinal block | 5 minutes after spinal block
  The investigators will measure cardiac output using non-invasive methods (USCOM) before spinal block and 5 minutes after spinal block.

SECONDARY OUTCOMES:
Total dose of vasopressor | 2 hours
  The investigators will record the total dose that treat hypotension during preoperative period
Number of patients who experience systolic blood pressure < 25% of preoperative measurement | 2 hours
  The investigators will monitor blood pressure at interval; before spinal block, then after spinal block every 1 minute for 10 for 10 times, every 2 minute for 5 times, every 3 minutes until delivery then every 5 minutes til the end of surgery. If the patient's systolic blood pressure is declined, vasopressor will be given.

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No